CLINICAL TRIAL: NCT00828620
Title: Imaging for Early Response Prediction to EGF-receptor Blocking Monoclonal Antibodies in Combination Therapy for Colorectal Cancer
Brief Title: Positron Emission Tomography - Computed Tomography (PET-CT) Cetuximab Project
Status: Terminated | Type: Observational
Why Stopped: Lack of recruitment
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s51276 - ML5241
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-06

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PET-CT: Patients with Unresectable stage IV colorectal cancer; eligible for 3rd line Irinotecan and Cetuximab
  Interventions: Other: Imaging study

INTERVENTIONS:
Other: Imaging study — PET-CT

SUMMARY:
Molecular imaging with positron emission tomography (PET) using [18F] fluorodeoxyglucose (FDG) has been suggested as an early, sensitive marker of tumour response to anticancer drugs by monitoring the changes in glucose metabolism in tumours. Recently, FDG-PET has shown to be highly sensitive in detecting early response in other tumours. In this study, the investigators will prospectively investigate the role of early FDG-PET (at day 7 and week 6) in outcome prediction.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven colorectal cancer
* Unresectable stage IV disease
* K-Ras wild type tumour
* Patients scheduled to undergo chemotherapy with irinotecan and cetuximab

Exclusion Criteria:

* Prior abdominal/pelvic radiotherapy, surgery or chemotherapy within 3 months prior to inclusion in the study
* Poorly controlled diabetes
* Concomitant serious illness, such as uncontrolled angina pectoris, myocardial infarction, heart failure, uncontrolled hypertension, infection
* Symptomatic brain metastases
* Pregnancy or participants of reproductive potential who are sexually active and not willing/able to use medically appropriate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: unresectable stage IV colorectal cancer pathologically proven measurable disease (RECIST) K-RAS wild type Eligible for 3rd line Irinotecan + Cetuximab Able for tolerate PET/CT imaging Serum glucose < 200mg/dl
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
PET response on day 7 | day 7

SECONDARY OUTCOMES:
To determine whether the PET criteria for response on day 7 correlates with the CT criteria of minimum 10% decrease in tumour size (RECIST) at week 6 | week 6
To define the optimal cutoff value of SUVmax and their predictive value | at day 7 and week 6
To explore the test/retest reliability of PET/CT in this setting | 2 weeks
To assess the value of PET/CT at day 7 in predicting overall survival | up to 1 year
To asses the correlations between biomarkers and PET changes after Cetuximab | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Cutsem, Prof.Dr, Principal Investigator — UZ Leuven
Locations (6):
- Belgium (6):
  - ZNA Middelheim, Antwerp
  - AZ Groeninge, Kortrijk
  - UZLeuven, Leuven
  - H Hart Roeselare Campus menen, Menen
  - Stedelijk Ziekenhuis Roeselare, Roeselare
  - Sint Augustinus Ziekenhuis, Wilrijk